CLINICAL TRIAL: NCT04667598
Title: Clinical and Metabonomics Study on the Treatment of Heart Failure After Myocardial Infarction With Modified Wenxin Decoction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jun Li (Other)
Responsible Party: Sponsor-Investigator, Jun Li, Li Jun, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JWWX-2020
Record Dates: First submitted 2020-11-23; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure; Myocardial Infarction
Keywords: Traditional Chinese Medicine
MeSH Terms: conditions — Heart Failure; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): On the basis of basic western medicine treatment (secondary prevention of coronary heart disease + anti-heart failure treatment), Patients in this group will be given modified Wenxin Tang granules, one dose per day, administered in two doses, 150-200 mL each time, for 12 weeks.
  Interventions: Drug: Modified Wenxin Decoction
- Control group (Placebo Comparator): On the basis of basic western medicine treatment (secondary prevention of coronary heart disease + anti-heart failure treatment), Patients in this group will be given placebo, one dose per day, administered in two doses, 150-200 mL each time, for 12 weeks.
  Interventions: Drug: Modified Wenxin Decoction

INTERVENTIONS:
Drug: Modified Wenxin Decoction — Mainly including make aconite , astragalus ， Cassia twig , dried ginger , red peony root , Chuanxiong , Codonopsis codonopsis , Ophiopogon ophiopogon , Schisandra , Stamen , Asarum , licorice.
  Other Names: placebo

SUMMARY:
To elucidate the efficacy and safety of weixin decoction in the treatment of heart failure after myocardial infarction.

DETAILED DESCRIPTION:
To elucidate the long-term protective effect of flavored Wenxin Decoction on heart failure after myocardial infarction.

To elucidate the effective components in the treatment of heart failure and the mechanism of metabolism regulation.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old；
* A history of acute myocardial infarction；
* Cardiac function Ⅱ - Ⅲ level；
* LVEF 50% or less;
* Nt-probnp level ≥ 450 pg/ mL；
* All men and women can sign the informed consent form.

Exclusion Criteria:

* Coronary artery bypass grafting was performed within 12 weeks；
* Undergo or possibly undergo cardiac resynchronization therapy;
* Primary valvular disease, left ventricular outflow tract obstruction, myocarditis, aneurysm, uncontrolled severe arrhythmia, cardiogenic shock, unstable angina pectoris, or acute myocardial infarction;
* Having a serious primary liver, kidney or blood system disease or having a serious mental illness or a systemic disease that is out of control;
* Serum creatinine > 194.5 mol/L or serum potassium > 5.5mmol /L;
* The level of alanine aminotransferase or alkaline phosphatase is 1.5 times of the normal upper limit of >;
* Abnormal blood pressure control, systolic blood pressure exceeding 180mmHg or diastolic blood pressure exceeding 110mmHg;
* Pregnancy or lactation; Known or suspected allergy to research drugs; To receive another investigational drug within 30 days of randomization or to be unwilling or unable to provide written consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Major cardiovascular events | One months after drug intervention
  Rates of cardiac death, acute myocardial infarction, stroke, and heart failure readmission

SECONDARY OUTCOMES:
Secondary indicators | Into the group day 1, week 4, week 8, week 12
  NT-proBNP， six-minute walking experiment and echocardiographic

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, MD, Study Director — Guang 'anmen Hospital of China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200
- [Result] Hildebrandt P. Systolic and nonsystolic heart failure: equally serious threats. JAMA. 2006 Nov 8;296(18):2259-60. doi: 10.1001/jama.296.18.2259. No abstract available. PMID 17090774
- [Result] Gheorghiade M, Bonow RO. Chronic heart failure in the United States: a manifestation of coronary artery disease. Circulation. 1998 Jan 27;97(3):282-9. doi: 10.1161/01.cir.97.3.282. No abstract available. PMID 9462531
- [Result] Gerber Y, Melton LJ 3rd, Weston SA, Roger VL. Association between myocardial infarction and fractures: an emerging phenomenon. Circulation. 2011 Jul 19;124(3):297-303. doi: 10.1161/CIRCULATIONAHA.110.007195. Epub 2011 Jun 27. PMID 21709062
- [Result] Ezekowitz JA, Kaul P, Bakal JA, Armstrong PW, Welsh RC, McAlister FA. Declining in-hospital mortality and increasing heart failure incidence in elderly patients with first myocardial infarction. J Am Coll Cardiol. 2009 Jan 6;53(1):13-20. doi: 10.1016/j.jacc.2008.08.067. PMID 19118718